CLINICAL TRIAL: NCT01403857
Title: Evaluating Liking, Acceptability and Health Benefits of Grain Products
Acronym: FL75
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WHNRC 235561-1
Record Dates: First submitted 2011-07-05; First posted 2011-07-27 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Food Preferences
Keywords: Acceptability; liking
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole Grain (Experimental): Whole grain products as defined by the American Association of Cereal Chemists (AACC) given in a market basket that contains eight commonly used grain products over six weeks.
  Interventions: Other: Whole grain foods
- Refined Grains (Placebo Comparator): Time control compared to experimental intervention.
  Interventions: Other: Refined grains

INTERVENTIONS:
Other: Whole grain foods — Eight commonly consumed whole grain products that meet the consumers Dietary Guidelines recommendations for a period of six weeks.
  Arms: Whole Grain
Other: Refined grains — Eight commonly consumed refined grain products given in amounts that fulfill the consumer's Dietary Guidelines for Americans recommendation over the course of six weeks.
  Arms: Refined Grains

SUMMARY:
The specific aims of the Grain Study are to determine if exposure to different types of grain products, over a period of 6 weeks, changes liking and acceptability and to determine if the gut microbiota, bacterial fermentation products, or gastrointestinal function changes with consumption of whole grains or refined grains.

DETAILED DESCRIPTION:
Subjects will be recruited in accordance with inclusion and exclusion criteria listed below. Subjects will be assigned to one of two different grain product 'exposure' groups - Group 1 will receive predominantly Whole Grain (WG) products and Group 2 will receive predominantly Refined Grain (RG) products (ratio of WG to RG assignment will be 2:1). For a 6-week exposure period, subjects will receive weekly market baskets of grain products consisting of breakfast cereals, breads, snack items, and side dishes with the target of providing whole grains at a level of 85% of grain intake for the WG group (this exceeds the current Dietary Guideline recommendation of 50%) and 15% for the RG group (this is the current estimated intake for U.S. adults). Before and after grain exposure, subjects will rate the acceptability and liking of numerous grain products. To accomplish this, subjects will participate in sensory evaluation tests using these products, and they will provide information using validated questionnaires and take implicit association tests. During the 6-week study period, subjects will record use of the market basket grain products, and provide subjective scores for taste, convenience, nutrition, and general liking. The quality of the total dietary intake will be assessed using unannounced 24-h recalls. Biological samples will also be collected from subjects. Blood and urine samples will be collected to evaluate risk factors of chronic disease, and biomarkers of whole grain intake, fruits and vegetables. Saliva and fecal samples will be collected to measure changes in gut microbiota and to measure metabolites of bacterial fermentation. Breath hydrogen tests will be conducted to measure bacterial fermentation. Two weeks after the end of the intervention period, subjects will participate in a nominal group session to identify significant barriers and facilitators to inclusion of grain products into their diets.

ELIGIBILITY:
Inclusion Criteria:

* 20-45 years of age
* male or female
* consumers of 1 or fewer whole grain products per day

Exclusion Criteria:

* Type I or II Diabetes or glucose intolerance
* Preference for whole grains
* Do not cook at home
* Pregnant or planning to be pregnant
* Smoking
* Chronic inflammatory bowel disease
* colorectal cancer
* Celiac disease or gluten sensitivity
* Crohn's disease
* Regular use of colonics and/or laxatives
* body weight change of >3% in last 6 months
* use of antibiotics, appetite suppressants, mood altering medications, and regular tobacco use.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2010-04; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in the acceptability and liking of grain products | 0, 6 weeks
  Sensory evaluation of grain products
Change in the gut microbiota and their fermentation products | 0, 6 weeks
  To determine if gut microbiota change over the intervention and if those changes persist over the long term. Gut microbiota assessed using 16S methodology.

SECONDARY OUTCOMES:
Change in gastrointestinal function | 0, 6 weeks
  Change in gastrointestinal function assessed using a questionnaire and exhaled breath hydrogen (ppm).
Liking the taste of grain products | 0, 6 weeks
  Implicit Attitude Tests assessed using a calculated D score using the method described by Greenwald et al.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Keim, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center; William Horn, MS, Study Director — USDA, Western Human Nutrition Research Center
Locations (1):
- Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Background] Greenwald AG, Nosek BA, Banaji MR. Understanding and using the implicit association test: I. An improved scoring algorithm. J Pers Soc Psychol. 2003 Aug;85(2):197-216. doi: 10.1037/0022-3514.85.2.197. PMID 12916565
- [Result] Cooper DN, Kable ME, Marco ML, De Leon A, Rust B, Baker JE, Horn W, Burnett D, Keim NL. The Effects of Moderate Whole Grain Consumption on Fasting Glucose and Lipids, Gastrointestinal Symptoms, and Microbiota. Nutrients. 2017 Feb 21;9(2):173. doi: 10.3390/nu9020173. PMID 28230784
- [Result] Cooper DN, Martin RJ, Keim NL. Does Whole Grain Consumption Alter Gut Microbiota and Satiety? Healthcare (Basel). 2015 May 29;3(2):364-92. doi: 10.3390/healthcare3020364. PMID 27417768
- [Result] De Leon A, Burnett DJ, Rust BM, Casperson SL, Horn WF, Keim NL. Liking and Acceptability of Whole Grains Increases with a 6-Week Exposure but Preferences for Foods Varying in Taste and Fat Content Are Not Altered: A Randomized Controlled Trial. Curr Dev Nutr. 2020 Mar 9;4(3):nzaa023. doi: 10.1093/cdn/nzaa023. eCollection 2020 Mar. PMID 32190809
- [Derived] De Leon A, Burnett DJ, Rust B, Lyly M, Keim NL. Initial implicit association between whole grains and taste does not predict consumption of whole grains in low-whole grain consumers: a pilot randomized controlled trial. Front Nutr. 2024 Sep 30;11:1408256. doi: 10.3389/fnut.2024.1408256. eCollection 2024. PMID 39403397